CLINICAL TRIAL: NCT06267027
Title: Comparison Of The Effects Of Kinesiotaping And High Intensity Laser Therapy In Patients With Lateral Epicondylitis: A Randomized Controlled Study
Brief Title: Comparison of Different Physical Therapy Modalities in Lateral Epicondylitis
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Bakirkoy Dr. Sadi Konuk Research and Training Hospital (Other Government)
Responsible Party: Principal Investigator, Sibel Caglar Okur, Principal Investigator, Bakirkoy Dr. Sadi Konuk Research and Training Hospital
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 2022/125
Record Dates: First submitted 2024-02-09; First posted 2024-02-20 (Actual); Last update posted 2024-02-20 (Actual); Status verified 2024-02

CONDITIONS: Lateral Epicondylitis
Keywords: Lateral epicondylitis; Kinesiotaping; High intensity laser
MeSH Terms: conditions — Tennis Elbow | interventions — Exercise

STUDY DESIGN:
Intervention Model Description: RANDOMIZED CONTROLLED STUDY
Who Masked: Investigator
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Exercise (Active Comparator): All study groups will be trained on a home exercise program that includes stretching and eccentric strengthening exercises.
  Interventions: Behavioral: Exercise
- Kinesiotaping and exercise (Experimental): This study groups will be trained on a home exercise program and kinesiotaping. Kinesiotaping, muscle inhibition and fascia correction techniques will be applied in the forearm as described by Kase et al.
  Interventions: Behavioral: Exercise; Device: Kinesiotaping
- High intensity laser therapy and exercise (Experimental): This study groups will be trained on a home exercise program and high intensity laser therapy.
  Interventions: Behavioral: Exercise; Device: High intensity laser therapy

INTERVENTIONS:
Behavioral: Exercise — The aim of exercise therapy is to stretch and strengthen the wrist extensor and flexor muscles. All study groups were given a home exercise program including stretching and eccentric strengthening exercises. The patient was instructed to start with stretching, and the patient was informed to stretch for 30s by flexing the wrist with the other hand while the shoulder was flexed 90 degrees, the elbow was in extension and the forearm was pronated. When stretching exercises could be performed painlessly, the patient was instructed to move on to strengthening exercises. Eccentric strengthening exercises for wrist extensors and flexors were explained with a support under the forearm and each patient was given a written program supported with visuals. It was emphasized that the exercises should be performed within the pain limit and patients were told to stop if they had severe pain. The exercise program was told to be performed 2 times a day, in 3 sets, 10 repetitions.
Device: Kinesiotaping — Area where the tape would be applied was clean and dry. If there is excessive hair in the application area, patients were asked to shave this area. It was explained that cream and similar substances should not be used. Muscle inhibition technique and fascia correction technique were used as the application technique. An X strip of approximately 25 cm and a Y strip of 10 cm in length are prepared as long as the distance between the lateral epicondyle and the wrist. The short arms of the X strip are adhered to the dorsal side of the hand without stretching and the crossed part of the strip is placed on the wrist with maximal stretching. The long arms of the X strip are adhered along the extensor carpi ulnaris and extensor carpi radialis to the lateral epicondyle without stretching. The Y strip was applied using the fascia correction method. The tails of the Y band were applied using an oscillating motion. The taping procedure was applied 2 times a week for 3 weeks for a total of 6 times.
  Arms: Kinesiotaping and exercise
Device: High intensity laser therapy — The elbow area was marked and then the epicondylitis protocol was selected. The epicondylitis protocol consists of 3 phases. Phase 1 and 2 consist of analgesic treatment and phase 3 consists of anti-inflammatory treatment. In phase 1 and phase 2 treatment protocol, 8 W was applied to a circular area with a radius of 1.0 cm for 3 min. In Phase 3 protocol, a dose of 80 J/cm2 at 8 W power was applied and the patient's treatment was completed.
  Arms: High intensity laser therapy and exercise

SUMMARY:
Comparison of the effects of kinesiotaping and high intensity laser therapy in patients with lateral epicondylitis: a randomized controlled study

DETAILED DESCRIPTION:
In this study, it was aimed to compare the effects of exercise therapy, kinesiology taping and high-intensity laser therapy on pain, muscle strength and functional status in patients with LE. Patients who applied to the outpatient clinic of the Sadi Konuk Training and Research Hospital Physical Medicine and Rehabilitation clinic due to elbow pain and were diagnosed with unilateral LE will be included. The study was planned as randomized, prospective and controlled. Patients will be randomized using a random (randomized) numbers table and distributed equally to the groups. Only exercise will be applied to the first group, high-intensity laser therapy and exercise to the second group, and kinesiology taping and exercise treatments to the third group. Sixty people will be included in the study. Patients will be evaluated before treatment, immediately after treatment, and at 4 weeks post-treatment. In the evaluation of the patients, the severity of pain during rest and activity measured with the Visual Analogue Scale (VAS), Quick Disability of the Arm, Shoulder and Hand (QuickDASH), Patient Based Lateral Epicondylitis Evaluation Test - Patient Rated Tennis Elbow Evaluation (PRTEE), Jamar' Hand grip strength will be evaluated with the hand dynamometer.

ELIGIBILITY:
Inclusion Criteria:

- Volunteer patients diagnosed with unilateral lateral epicondylitis

Exclusion Criteria:

* Those who have previously received treatment for lateral epicondylitis
* Current extremity fracture or surgical history
* Presence of congenital deformity in the upper extremity
* Cervical radiculopathy, myelopathy, plexopathy, entrapment neuropathies
* Presence of neurological disease such as stroke, Parkinson's, multiple sclerosis, epilepsy and muscle disease
* Presence of skin lesion, infection and open wound on the affected extremity
* Presence of metal implant in the affected extremity
* Rheumatological disease
* Pregnancy
* Pacemaker presence
* Malignancy
* Cognitive dysfunction
* Presence of psychiatric illness

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 55 (Actual)
Dates: Start 2023-02-07 (Actual); Primary Completion 2023-09-15 (Actual); Study Completion 2023-12-15 (Actual)

PRIMARY OUTCOMES:
Patient Rated Tennis Elbow Evaluation (PRTEE) | Initial, Week 3, Week 7
  It consists of pain and function subscales that assess the level of pain in the affected arm in the last 1 week and the degree of difficulty experienced during specific and daily activities. The pain assessment consists of 5 questions and the functional assessment consists of 10 questions, totaling 15 questions. The questions are evaluated with a 10-point Likert scale, as in the VAS, with numbers written side by side from 0 to 10. It is calculated by averaging the pain score and functional score. The total score ranges from 0-100, with a higher score indicating an increase in pain and functional loss. Validation of turkish version is available.

SECONDARY OUTCOMES:
Visual Analogue Scale (VAS) | Initial, Week 3, Week 7
  The VAS is a simple, subjective measurement method used to assess the patient's pain intensity and response to treatment. On a 10 cm chart, patients are asked to indicate the severity of their pain within 24 hours, with 0 representing no pain and 10 representing unbearable pain.
Quick Disabilities of the Arm, Shoulder and Hand (qDASH) | Initial, Week 3, Week 7
  Quick-DASH is a shortened version of the 30-question DASH questionnaire used to assess participation and activity limitations in upper extremity musculoskeletal disorders. Patients strain during activities of daily living in the past week is assessed with 11 questions. Answers are scored from 1 to 5 on a scale from good to bad (1: no difficulty, 2: mild difficulty, 3: moderate difficulty, 4: extreme difficulty, 5: unable to do at all). The total score ranges from 0-100. Validation of turkish version is available.
Jamar's handheld dynamometer | Initial, Week 3, Week 7
  Hand grip strength was evaluated with the Jamar hand dynamometer recommended by the American Society for Surgery of the Hand. The recommended hand grip strength measurement was evaluated with the patient in a sitting position, shoulder in adduction and neutral rotation, elbow in 90 degree flexion, forearm and wrist in neutral position. The patient's grip strength until the onset of pain is used for measurement. Three measurements are made with a one-minute interval between each measurement and averaged. All measurements were performed in both hands, first on the pain-free arm and then on the side with LE.

CONTACTS AND LOCATIONS:
Overall Officials: Sibel CAGLAR, Principal Investigator — Bakırkoy Dr. Sadi Konuk Training and Research Hospital; Hasan YUKSEL, Study Chair — Bakırkoy Dr. Sadi Konuk Training and Research Hospital
Locations (1):
- BakirkoySadiKonuk, Bakırköy, Istanbul, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Cho YT, Hsu WY, Lin LF, Lin YN. Kinesio taping reduces elbow pain during resisted wrist extension in patients with chronic lateral epicondylitis: a randomized, double-blinded, cross-over study. BMC Musculoskelet Disord. 2018 Jun 19;19(1):193. doi: 10.1186/s12891-018-2118-3. PMID 29921250
- [Background] Kaydok E, Ordahan B, Solum S, Karahan AY. Short-term Efficacy Comparison of High-intensity and Low-intensity Laser Therapy in the Treatment of Lateral Epicondylitis: A Randomized Double-blind Clinical Study. Arch Rheumatol. 2019 Apr 24;35(1):60-67. doi: 10.5606/ArchRheumatol.2020.7347. eCollection 2020 Mar. PMID 32637921
- [Background] Shechtman O, Gestewitz L, Kimble C. Reliability and validity of the DynEx dynamometer. J Hand Ther. 2005 Jul-Sep;18(3):339-47. doi: 10.1197/j.jht.2005.04.002. PMID 16059855
- [Background] Haidar SG, Kumar D, Bassi RS, Deshmukh SC. Average versus maximum grip strength: which is more consistent? J Hand Surg Br. 2004 Feb;29(1):82-4. doi: 10.1016/j.jhsb.2003.09.012. PMID 14734079
- [Background] Halpern CA, Fernandez JE. The effect of wrist and arm postures on peak pinch strength. J Hum Ergol (Tokyo). 1996 Dec;25(2):115-30. PMID 9735592
- [Background] Angst F, Schwyzer HK, Aeschlimann A, Simmen BR, Goldhahn J. Measures of adult shoulder function: Disabilities of the Arm, Shoulder, and Hand Questionnaire (DASH) and its short version (QuickDASH), Shoulder Pain and Disability Index (SPADI), American Shoulder and Elbow Surgeons (ASES) Society standardized shoulder assessment form, Constant (Murley) Score (CS), Simple Shoulder Test (SST), Oxford Shoulder Score (OSS), Shoulder Disability Questionnaire (SDQ), and Western Ontario Shoulder Instability Index (WOSI). Arthritis Care Res (Hoboken). 2011 Nov;63 Suppl 11:S174-88. doi: 10.1002/acr.20630. No abstract available. PMID 22588743
- [Background] Overend TJ, Wuori-Fearn JL, Kramer JF, MacDermid JC. Reliability of a patient-rated forearm evaluation questionnaire for patients with lateral epicondylitis. J Hand Ther. 1999 Jan-Mar;12(1):31-7. doi: 10.1016/s0894-1130(99)80031-3. PMID 10192633
- [Background] Altan L, Ercan I, Konur S. Reliability and validity of Turkish version of the patient rated tennis elbow evaluation. Rheumatol Int. 2010 Jun;30(8):1049-54. doi: 10.1007/s00296-009-1101-6. Epub 2009 Aug 26. PMID 19707766